CLINICAL TRIAL: NCT02528344
Title: The Effects of High-Intensity Interval Training on Inflammation in Adults With Rheumatoid Arthritis
Brief Title: High Intensity Interval Training and Rheumatoid Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00064057
Record Dates: First submitted 2015-08-17; First posted 2015-08-19 (Estimated); Last update posted 2016-12-08 (Estimated); Status verified 2016-06

CONDITIONS: Rheumatoid Arthritis
Keywords: High Intensity Interval Training
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HIIT - RA (Experimental): All participants will undergo high intensity interval training 3x/week for 10-12 weeks. Intense exercise will be interspersed with appropriate rest periods of low intensity exercise
  Interventions: Behavioral: HIIT

INTERVENTIONS:
Behavioral: HIIT — All participants will undergo high intensity interval training 3x/week for 10-12 weeks. Intense exercise will be interspersed with appropriate rest periods of low intensity exercise

SUMMARY:
The overall objective is to determine whether High Intensity Interval Training (HIIT) has potential to improve disease activity scores for Rheumatoid Arthritis (RA) patients. By reducing inflammation and modifying immune function HIIT may offer a substantial paradigm shift in RA care, especially in older persons with RA who experience aging related-immunesenescence, increased systemic inflammation and greater physical inactivity than young persons. Prior to embarking on a large scale trial of HIIT-induced disease modification, this pilot study aims to demonstrate that HIIT can produce measurable responses in disease activity scores and peak VO2in persons undergoing routine pharmacologic treatment for RA.

ELIGIBILITY:
Inclusion Criteria:

* Seropositive (positive rheumatoid factor or anti-citrullinated protein antibody) or erosions typical of RA on radiographs.
* History of fulfilling 2010 ACR/EULAR Classification Criteria for RA
* Able to walk on a treadmill
* Not participating in regular physical exercise (more than 60 minutes of moderate intensity or 30 minutes of vigorous intensity exercise per week) or weight reduction dieting.
* No medication changes within the last three months.
* Willing to forego knee joint injections, regular NSAID use, and use acetaminophen for any necessary analgesia during the course of the intervention.
* No current (within the last three weeks) pharmacologic therapy with corticosteroids.

Exclusion Criteria:

* Coronary artery disease
* Diabetes mellitus
* Chronic obstructive pulmonary disease
* Absolute contra-indications to exercise: Recent (<6 months) acute cardiac event unstable angina, uncontrolled dysrhythmias causing symptoms or hemodynamic compromise, symptomatic aortic stenosis, uncontrolled symptomatic heart failure, acute pulmonary embolus, acute myocarditis or pericarditis, suspected or known dissecting aneurism and acute systemic infection.
* Other inflammatory arthropathy or myopathy, Paget's disease, pigmented villonodular synovitis, joint infection, ochronosis, neuropathic arthropathy, osteochondromatosis, acromegaly, hemochromatosis, Wilson's disease, osteonecrosis, knee replacement.
* Contraindicated Medicine: ticlopidine, clopidogrel, dipyridamole, warfarin, heparin, enoxaparin and other blood thinners.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2015-09; Primary Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Change in Disease Activity Scores | Baseline and Post-Intervention (12-weeks)

SECONDARY OUTCOMES:
Change in Peak Oxygen Consumption | Baseline and Post-Intervention (12-weeks)

CONTACTS AND LOCATIONS:
Locations (1):
- Duke Molecular Physiology Institute, Durham, North Carolina, United States

REFERENCES:
- [Derived] Andonian BJ, Koss A, Koves TR, Hauser ER, Hubal MJ, Pober DM, Lord JM, MacIver NJ, St Clair EW, Muoio DM, Kraus WE, Bartlett DB, Huffman KM. Rheumatoid arthritis T cell and muscle oxidative metabolism associate with exercise-induced changes in cardiorespiratory fitness. Sci Rep. 2022 May 6;12(1):7450. doi: 10.1038/s41598-022-11458-4. PMID 35523821
- [Derived] Andonian BJ, Johannemann A, Hubal MJ, Pober DM, Koss A, Kraus WE, Bartlett DB, Huffman KM. Altered skeletal muscle metabolic pathways, age, systemic inflammation, and low cardiorespiratory fitness associate with improvements in disease activity following high-intensity interval training in persons with rheumatoid arthritis. Arthritis Res Ther. 2021 Jul 10;23(1):187. doi: 10.1186/s13075-021-02570-3. PMID 34246305
- [Derived] Andonian BJ, Bartlett DB, Huebner JL, Willis L, Hoselton A, Kraus VB, Kraus WE, Huffman KM. Effect of high-intensity interval training on muscle remodeling in rheumatoid arthritis compared to prediabetes. Arthritis Res Ther. 2018 Dec 27;20(1):283. doi: 10.1186/s13075-018-1786-6. PMID 30587230
- [Derived] Bartlett DB, Willis LH, Slentz CA, Hoselton A, Kelly L, Huebner JL, Kraus VB, Moss J, Muehlbauer MJ, Spielmann G, Kraus WE, Lord JM, Huffman KM. Ten weeks of high-intensity interval walk training is associated with reduced disease activity and improved innate immune function in older adults with rheumatoid arthritis: a pilot study. Arthritis Res Ther. 2018 Jun 14;20(1):127. doi: 10.1186/s13075-018-1624-x. PMID 29898765